CLINICAL TRIAL: NCT04462614
Title: Feasibility to Stop Perdialytic Heparin Therapy in Hemodialysed Patients With HeprAN ™ Membrane and Treated by Long-term Anticoagulation With VKA
Brief Title: Possibility to Stop Perdialytic Heparin Therapy in Hemodialysed Patients With HeprAN ™ Membrane and Treated by Long-term Anticoagulation With VKA
Acronym: REMARK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PO20091
Record Dates: First submitted 2020-07-03; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Chronic Hemolysis; VKA; Anticoagulants / Administration & Dosage; Coated Materials; Biocompatible; Heparin / Administration & Dosage; Membranes Artificial; Prospective Studies; Renal Dialysis / Methods; Renal Insufficiency / Therapy
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single-arm study (Experimental): Chronic hemodialysis patients for at least 3 months at Reims University Hospital, treated by long-term anticoagulation with VKA and dialysed with the HeprAN ™ membrane
  Interventions: Drug: Decrease per-dialytic heparin therapy

INTERVENTIONS:
Drug: Decrease per-dialytic heparin therapy — Week 1: maintenance's dose stop Week 2: 50% drop in the loading dose Week 3: complete cessation of heparin therapy during the session.

SUMMARY:
Use HeprAN ™ membrane (coated with heparin) should be allow the success of dialysis sessions, with adequate dialysis parameters, in patients treated by long-term anticoagulation with VKA, without addition of heparin perdialytic.

Less use of heparin (UFH or LMWH) during hemodialysis session should be allow a decrease of bleedings (moderate or major) and blood transfusions for hemodialysed patients with HeprAN ™ membrane and treated by long-term anticoagulation with VKA

DETAILED DESCRIPTION:
The aim will be to study possibility of hemodialysis sessions success, without perdialytic anticoagulation but with adequate dialysis parameters (defined by the patient's Kt / V machine), in patients treated by long-term anticoagulation with VKA and dialysed with the HeprAN ™ membrane.

ELIGIBILITY:
inclusion criteria :

* 18 years old and older
* chronic hemodialysis for at least 3 months
* treated by long-term anticoagulation with VKA
* hemodialysis with the HeprAN® membrane
* per dialytic heparin therapy (UFH or LMWH)
* dialyzed at Reims University Hospital
* agreeing to participate in the study

Exclusion criteria

* chronic hemodialysis without per dialytic heparin
* Patient dialized with single lumen catheter for vascular access
* less than 18 years old
* pregnant or lactating women
* protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Failure of heparin withdrawal in patients treated by long-term anticoagulation with VKA and dialysed with the HeprAN ™ membrane, verify adequate dialysis parameters | 3 weeks
  Failure is defined by
  * early interruption of the dialysis session (<95% of the prescribed time) for :
  * extracorporeal circuit coagulation
  * recurrent venous pressure alarm causing blood pump shutdown or
  * Lower quality of dialysis compared to the quality before stopping perdialytic anticoagulation (defined as Kt/V less than - 2SD for 3 consecutive sessions)

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France